CLINICAL TRIAL: NCT02521207
Title: A Two-Part, Randomised, Open-Label, Evaluator-Blinded, Multiple-Dose, Phase I Pilot Study With OXP001 Ibuprofen 400 mg Tablets and Brufen® 400 mg Tablets to Assess the Comparative Bioavailability (Part 1) and Effects on Gastroduodenal Irritation (Part 2) in Healthy Human Subjects
Brief Title: Pilot Study of OXP001(2) and Brufen in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oxford Pharmascience Ltd (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OXP001-003
Record Dates: First submitted 2015-08-05; First posted 2015-08-13 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Gastroduodenal Erosions
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part 1 OXP001 (Experimental): OXP001 formulation containing 800mg ibuprofen single dose
  Interventions: Drug: Ibuprofen
- Part 1 Ibuprofen control (Active Comparator): Ibuprofen control 800mg single dose
  Interventions: Drug: Ibuprofen
- Part 2 OXP001 (Experimental): OXP001 formulation containing 800mg ibuprofen three times per day
  Interventions: Drug: Ibuprofen
- Part 2 Ibuprofen control (Experimental): Ibuprofen control 800mg three times per day
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen

SUMMARY:
The study will compare the study drug to an already marketed formulation of prescription strength ibuprofen (Brufen® the reference product) by looking at how the drug is taken up by the body and also by performing a specialist procedure called an endoscopy (or more specifically, a gastroscopy). The safety and tolerability of the study drug will also be assessed.

The study will consist of 2 parts involving up to 54 healthy male and female subjects. Subjects will be randomly assigned to receive either the study drug or reference product. Part 1 will be a cross over study in which up to 10 subjects will receive a single dose of 800 mg study drug OXP001 or Brufen® on Day 1, then a single dose of 800 mg study drug OXP001 or Brufen® on Day 4. Part 1 will assess bioavailability and involve an interim decision on progression to Part 2. In Part 2, up to 44 subjects will receive a dose of 800 mg OXP001 or Brufen® three times daily for 7 days in order to assess pharmacokinetics and stomach irritation using endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subject
* Healthy, normal upper GI tract as indicated by no ulcers or erosions at baseline, as assessed by the gastroenterologist conducting the endoscopy (ie Lanza score of 0 in both the stomach and duodenum) (Part 2 only)
* H. pylori negative

Exclusion Criteria:

* Clinically significant abnormal laboratory parameters
* Any clinically significant diseases or conditions affecting the haematopoietic, cardiovascular, renal, hepatic, endocrine, pulmonary, central nervous, immunological, dermatological, GI or any other body system

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Part 1: Comparison of Peak Plasma Concentration (Cmax) | Part 1; Day 1 and Day 4
Part 2: Comparison of Average Lanza Score | Part 2; Day 8
Part 2: Comparison of Average Number of Erosions | Day 8
Part 1: Comparison of Area Under the Curve (AUC) | Part 1; Day 1 and Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mair, Principal Investigator — Quotient Clinical Ltd
Locations (1):
- Quotient Clinical Ltd, Nottingham, Notts, United Kingdom